CLINICAL TRIAL: NCT03917888
Title: Clinical Impact of Lung Ultrasound Monitoring for Diagnosis of Ventilator Associated Pneumonia: a Diagnostic Randomized Controlled Trial.
Brief Title: Clinical Impact of Lung Ultrasound Monitoring for Diagnosis of VAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Saurabh Pradhan, MD, DM (Critical care medicine), Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 78611
Record Dates: First submitted 2019-04-10; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Ventilator Associated Pneumonia
Keywords: ventilator associated pneumonia; lung ultrasound
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung ultrasound (Experimental): Patients will be monitored for ventilator associated pneumonia using lung ultrasound combined with clinical features
  Interventions: Diagnostic Test: lung ultrasound
- Chest x-ray (No Intervention): Patients will be monitored for ventilator associated pneumonia using chest x-ray and clinical features.

INTERVENTIONS:
Diagnostic Test: lung ultrasound — lung ultrasound will be performed daily in mechanically ventilated patients after 48 hours of ventilation to screen for ventilator associated pneumonia
  Arms: Lung ultrasound

SUMMARY:
The study evaluates whether lung ultrasound monitoring could lead to earlier detection of ventilator associated pneumonia and influence outcome. Half of the participants will be diagnosed with VAP using a combination of lung ultrasound and clinical features and half will be diagnosed using the Johanson criteria, which is a combination of clinical features and chest x-ray.

DETAILED DESCRIPTION:
The current guidelines recommend the use of chest x-ray or computed tomography of the chest to aid in the diagnosis of VAP. However many studies have shown that chest x-ray is neither very sensitive nor specific for pneumonia, and computed tomography, though has the highest diagnostic accuracy, is not routinely performed due to logistics, safety concerns, economics and radiation exposure.

Emerging studies including meta-analyses have shown high sensitivity and specificity of lung ultrasound in diagnosing pneumonia. When combined with clinical and microbiological features it has shown to be helpful in early diagnosis of VAP, but a study to show whether such early detection improves outcome is lacking.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation for more than 48 hours
* Absence of pneumonia as the reason for mechanical ventilation (includes clinical, radiological or sonographic diagnosis)

Exclusion Criteria:

* Recent trauma or surgery to the thorax (including chest tube insertion)
* Presence of dressings or skin conditions restricting access to the thorax
* Confirmed pregnancy
* If already enrolled in the study
* Denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
ventilator free days | day 28 from diagnosis of VAP
  number of days alive from day 1 (of VAP) to day 28 on which a patient breathes without assistance, if the period of unassisted breathing lasted at least 48 consecutive hours. If death occurs within 28 days then ventilator free days is counted as 0

SECONDARY OUTCOMES:
icu mortality | through study completion, an average of 3 months
  death during icu stay
icu length of stay | through study completion, an average of 3 months
  total duration of stay in icu
delta sofa | day 4 from VAP diagnosis
  change in Sequential Organ Failure Score (SOFA) at day 4 of onset of VAP from the day of onset of VAP. SOFA ranges from 0 to 24. Delta sofa is the difference between SOFA score at day 4 from day 0 of VAP diagnosis. the higher the difference, the better the outcome
ventilator days | day 28 from intubation
  total days the patient remains in mechanical ventilation
antibiotic duration | day 14 from initiation of antibiotic
  total days the patient receives antibiotics for VAP

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Pradhan, DM, Principal Investigator — Institute of Medicine, TUTH
Locations (1):
- Tribhuvan university teaching hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
all data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: access will be shared on request